CLINICAL TRIAL: NCT02740985
Title: A Phase 1, Open-Label, Multicenter Study to Assess Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-Tumor Activity of Ascending Doses of AZD4635 Both as Monotherapy and in Combination in Patients With Advanced Solid Malignancies
Brief Title: A Phase 1 Clinical Study of AZD4635 in Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8730C00001; REFMAL 435 (Other: Sarah Cannon Development Innovations, LLC)
Record Dates: First submitted 2016-02-29; First posted 2016-04-18 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Advanced Solid Malignancies; Non-Small Cell Lung Cancer (NSCLC); Metastatic Castrate-Resistant Prostate Carcinoma (mCRPC); Colorectal Carcinoma (CRC)
Keywords: AZD4635; durvalumab; oleclumab; docetaxel; non-small cell lung cancer; advanced solid malignancies; prostate cancer; colorectal cancer; abiraterone acetate; enzalutamide
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Prostatic Neoplasms | interventions — durvalumab; Abiraterone Acetate; enzalutamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- Arm A (Experimental): AZD4635 monotherapy as nanoparticle suspension 125 mg BID
  Interventions: Drug: AZD4635
- Arm B (Experimental): AZD4635 monotherapy as nanoparticle suspension 75 mg QD
  Interventions: Drug: AZD4635
- Arm C (Experimental): AZD4635 monotherapy as nanoparticle suspension 100 mg QD
  Interventions: Drug: AZD4635
- Arm D (Experimental): AZD4635 as nanoparticle suspension 75 mg QD plus durvalumab
  Interventions: Drug: AZD4635; Drug: Durvalumab
- Arm E (Experimental): AZD4635 as nanoparticle suspension 100 mg QD plus durvalumab
  Interventions: Drug: AZD4635; Drug: Durvalumab
- Arm EA (Experimental): AZD4635 as nanoparticle suspension plus enzalutamide
  Interventions: Drug: AZD4635; Drug: Enzalutamide
- Arm AA (Experimental): AZD4635 as nanoparticle suspension plus abiraterone acetate
  Interventions: Drug: AZD4635; Drug: Abiraterone Acetate
- Arm F (Experimental): AZD4635 as nanoparticle suspension plus durvaluamb in patients post immunotherapy with non-small cell lung cancer. Patients will be allocated randomly (1:1) between Arms F and G.
  Interventions: Drug: AZD4635; Drug: Durvalumab
- Arm G (Experimental): AZD4635 monotherapy as nanoparticle suspension in patients post immunotherapy with non-small cell lung cancer. Patients will be allocated randomly (1:1) between Arms F and G.
  Interventions: Drug: AZD4635
- Arm H (Experimental): AZD4635 monotherapy as nanoparticle suspension in patients post immunotherapy with other solid tumours.
  Interventions: Drug: AZD4635
- Arm I (Experimental): AZD4635 as nanoparticle suspension plus durvalumab in immunotherapy naïve patients with metastatic castration resistant prostate cancer. Patients will be allocated randomly (1:1) between Arms I and J.
  Interventions: Drug: AZD4635; Drug: Durvalumab
- Arm J (Experimental): AZD4635 monotherapy as nanoparticle suspension in immunotherapy naïve patients with metastatic castration resistant prostate cancer. Patients will be allocated randomly (1:1) between Arms I and J.
  Interventions: Drug: AZD4635
- Arm K (Experimental): AZD4635 monotherapy as nanoparticle suspension in immunotherapy naïve patients with colorectal carcinoma.
  Interventions: Drug: AZD4635
- Arm KD (Experimental): AZD4635 as nanoparticle suspension plus durvalumab in immunotherapy-naïve patients with colorectal carcinoma.
  Interventions: Drug: AZD4635; Drug: Durvalumab
- Arm L (Experimental): AZD4635 monotherapy as nanoparticle suspension in immunotherapy naïve patients with other solid tumours.
  Interventions: Drug: AZD4635
- Arm CA (Experimental): AZD4635 capsule formulation monotherapy 75 mg, 150 mg, and 200 mg QD. A lower dose of 125 mg or 100 mg may be given. The pharmacokinetics of the single dose AZD4635 capsule formulation will be characterized on Cycle 1 Day 1 in Arm CA. Steady-state pharmacokinetics will be assessed on Cycle 1 Day 15. Cycle 1 and Cycle 2 will be administered in 3-week cycles to assess the safety and dose-limiting toxicity (DLT). After Cycle 1, PKs will be collected on Day 1 of every even numbered cycle (Cycles 2, 4, and 6).
  Interventions: Drug: AZD4635
- Arm CB (Experimental): AZD4635 capsule formulation 50 mg QD or 75 mg QD plus durvalumab and oleclumab. The pharmacokinetics of AZD4635 capsule formulation will be characterized on Cycle 1, 2, and 4 (Day 1) in Arm CB. Steady-state pharmacokinetics will be assessed on Cycle 2 Day 15. Cycle 1 will be administered in a 3-week cycle to assess the safety and dose-limiting toxicity (DLT). PKs will also be collected on Day 1 of Cycles 3 and 5.
  Interventions: Drug: AZD4635; Drug: Durvalumab; Drug: Oleclumab
- Arm CC (Experimental): AZD4635 capsule formulation 50 mg QD or 75 mg QD plus docetaxel. The pharmacokinetics of the single dose AZD4635 capsule formulation will be characterized on Cycle 1 Day 1 in Arm CC. Steady-state pharmacokinetics will be assessed on Cycle 1 Day 15. Cycles will be administered in 3-week cycles to assess the safety and dose-limiting toxicity (DLT). After Cycle 1, PKs will be collected on Day 1 of every even numbered cycle (Cycles 2, 4, and 6).
  Interventions: Drug: AZD4635; Drug: Docetaxel

INTERVENTIONS:
Drug: AZD4635 — AZD4635 will be administered orally as a nanosuspension or capsule on a continuous schedule in Arms A, B, C, D, E, F, G, H, I, J, K, KD, L, AA, and EA. The AZD4635 nanoparticle drug product will be constituted extemporaneously as an oral suspension by the patient immediately prior to dosing. In Arms CA, CB, and CC AZD4635 will be administered as 75 mg or 50 mg capsules. Additionally, in Arm CA, AZD4635 will also be administered at 150 mg and 200 mg, or a lower dose of 125 mg or 100 mg may be given.
Drug: Durvalumab — Durvalumab will be administered by intravenous infusion once every 4 weeks. Durvalumab should be reconstituted using aseptic techniques with sterile water for injection. The reconstituted solution will be diluted with 0.9% (w/v) saline prior to IV infusion.
  Other Names: MEDI4736
  Arms: Arm CB; Arm D; Arm E; Arm F; Arm I; Arm KD
Drug: Abiraterone Acetate — Abiraterone acetate 1000 mg PO QD will be given with prednisone BID. The patient must receive abiraterone/prednisone according to the prescribing information during the DLT assessment period, Cycle 1 and Cycle 2. After Cycle 2 necessary abiraterone/ prednisone dose modifications may follow institutional standard practice.
  Abiraterone acetate is supplied in 250 mg tablets.
  Other Names: Zytiga
  Arms: Arm AA
Drug: Enzalutamide — Enzalutamide 160 mg PO QD will be dosed per the approved package insert. The patient must receive enzalutamide according to the prescribing information during the DLT assessment period, Cycle 1 and Cycle 2. After Cycle 2 necessary enzalutamide dose modifications may follow institutional standard practice.
  Enzalutamide is supplied as 40 mg soft gelatin capsules.
  Other Names: Xtandi
  Arms: Arm EA
Drug: Oleclumab — Oleclumab 1500 mg will be given by IV infusion on Days 1 and 15 of each cycle.
  Other Names: MEDI9447
  Arms: Arm CB
Drug: Docetaxel — Patients in Cohort CC will receive docetaxel 75 mg/m² by IV infusion according to institutional standards of practice on Day 1 of each treatment cycle. If a patient's body surface area is greater than 2.2 m², the docetaxel dose will be adjusted to a body surface area of 2.2 m².
  The patient should be pre-medicated with oral dexamethasone 8 mg (or equivalent) twice daily starting the day prior to treatment for a total of 3 days, or according to institutional standards of practice.
  Other Names: Taxotere
  Arms: Arm CC

SUMMARY:
This is a Phase 1, open-label, multicenter study of continuous oral dosing of AZD4635 administered to patients with advanced solid malignancies. Dosing will be escalated until a maximum-tolerated dose (MTD) is determined in patients. The MTD will be defined by dose-limiting toxicity. The study design allows an escalation of dose with intensive safety monitoring to ensure the safety of the patients. Expansion cohorts will further assess safety and preliminary anti-tumor activity in a variety of advanced solid tumor malignancies. Other dosing schedules and/or combinations may be evaluated based on the emerging PK and safety data.

The primary objectives of this study are to:

* Investigate the safety and tolerability of AZD4635 monotherapy when given orally (PO) to patients with advanced solid malignancies.
* Investigate the safety, tolerability, and pharmacokinetics (PK) of AZD4635 monotherapy capsule formulation when given to patients with advanced solid malignancies.
* Investigate the safety and tolerability of AZD4635 PO when given in combination with durvalumab, durvalumab plus oleclumab, or docetaxel to patients with advanced solid malignancies and to investigate the safety and tolerability of AZD4635 in combination with abiraterone acetate or enzalutamide in patients with mCRPC.
* Define the maximum-tolerated dose (MTD) of AZD4635 in combination with durvalumab.
* Define the recommended Phase 2 dose (RP2D) of AZD4635 in combination with abiraterone acetate or enzalutamide.
* Determine the safety, tolerability, and immune effects of AZD4635 when administered in combination with durvalumab to patients with non-small cell lung cancer (NSCLC) who have previously received immunotherapy (Phase 1b portion).
* Investigate the safety and tolerability of AZD4635 capsule formulation in combination with durvalumab and oleclumab when given to patients with mCRPC or advanced solid tumor malignancy.
* Define the RP2D of AZD4635 capsule formulation in combination with durvalumab and oleclumab when given to patients with mCRPC or advanced solid tumor malignancy.
* Investigate the safety and tolerability of AZD4635 capsule formulation in combination with docetaxel when given to patients with mCRPC or advanced solid tumor malignancy.
* Define the RP2D of AZD4635 capsule formulation in combination with docetaxel when given to patients with mCRPC or advanced solid tumor malignancy.

DETAILED DESCRIPTION:
The study will be conducted in two segments. The first segment of the study, designated Phase 1a, will be a dose escalation design in order to assess the safety, tolerability, pharmacokinetics (PK), and preliminary anti-tumor activity of ascending doses of AZD4635 as monotherapy, in combination with durvalumab or durvalumab plus oleclumab, in combination with docetaxel, and in combination with either abiraterone acetate or with enzalutamide.

A capsule formulation of AZD4635 will be evaluated in 3 arms (arms CA, CB, and CC). An oral nanoparticle suspension in water constituted extemporaneously by the patient will be administered in all other treatment arms. Most patients who started therapy with the nanoparticle suspension will transition to the capsule dosage form depending on the arm they are assigned to and emerging data. Active patients in arms C, D, E, F, G, H, I, J, K, KD, and L should be offered the option to transition to the capsule formulation at the discretion of the Investigator in discussion with the Medical Monitor. Patients in study arms AA and AE receiving AZD4635 as the nanoparticle suspension should change over to the capsule formulation as soon as possible at the discretion of the Investigator.

The dose escalation arms are described as follows:

* Arms A, B, and C (dose escalation of AZD4635 monotherapy).
* Arms CA, CB, and CC. In arm CA, the safety, tolerability and PK of the capsule formulation will be assessed in approximately 6 patients with advanced solid malignancies to ensure at least 5 patients have evaluable pharmacokinetic sampling. An additional 12 patients will be enrolled in this arm. Arm CB will assess the safety and tolerability and determine the RP2D of the AZD4635 capsule plus durvalumab and oleclumab in approximately 12 patients. Arm CC will assess the safety, tolerability and determine the RP2D of AZD4635 capsule plus docetaxel in approximately 12 patients .
* Arms D and E [dose escalation of AZD4635 in combination with durvalumab anti-programmed death-ligand 1 (PD-L1)].

Arms A through E enrolled 38 patients in Phase 1a in order to establish the Recommended Phase 2 Dose (RP2D) of the nanoparticle suspension formulation of AZD4635 as a single agent or in combination with durvalumab.

● Arms EA and AA. Arms EA and AA [dose escalation of AZD4635 in combination with either abiraterone acetate plus prednisone or enzalutamide in patients with metastatic castrate-resistant prostate cancer (mRCPC)]. The AZD4635 plus hormonal therapy cohorts will enroll concurrently. Patients who previously received abiraterone acetate, enzalutamide, or apalutamide as part of their prior treatments for mCRPC may be enrolled to the enzalutamide plus AZD4635 arm (Cohort EA) or the abiraterone acetate plus AZD4635 arm (Cohort AA) at the discretion of the Investigator. Approximately 24 to 48 patients with mCRPC will be treated in the AZD4635 plus hormonal therapy arms in order to establish the RP2D.

In Phase 1a approximately 90-132 patients will be treated with AZD4635 as a single agent or in combination with durvalumab, durvalumab plus oleclumab, docetaxel, abiraterone acetate or enzalutamide.

The second segment of the study, designated Phase 1b, will further assess the safety and preliminary activity in the expansion arms described below.

* Arm F - AZD4635 in combination with durvalumab. Post-immunotherapy non-small cell lung cancer (NSCLC). [15 patients]
* Arm G - AZD4635 monotherapy. Post-immunotherapy NSCLC. [15 patients]
* Arm H - AZD4635 monotherapy. Immune checkpoint resistant malignancies, previously treated with approved immunotherapy and progressed or responded and then stopped responding (e.g. renal cell carcinoma, head and neck carcinoma, or MSI high cancers which have approved settings for anti-PD-1 treatment).[20 patients]
* Arm I - AZD4635 in combination with durvalumab. Immune checkpoint naïve mCRPC.[40 patients]
* Arm J - AZD4635 monotherapy. Immune checkpoint naïve CRPC. [40 patients]
* Arm K - AZD4635 monotherapy. Immune checkpoint naïve colorectal carcinoma (CRC). CRC, excluding MSI high, which has not been treated with immune checkpoint inhibitors. [20 patients]
* Arm KD - AZD4635 in combination with durvalumab. Immune checkpoint naïve CRC. CRC, excluding MSI high, which has not been treated with immune checkpoint inhibitors. [20 patients]
* Arm L - AZD4635 monotherapy. Other solid tumours immune checkpoint naïve. Relapsed/refractory tumors which have not been treated with immune checkpoint inhibitors. [20 patients]

Patients will be randomly assigned between open-label arms with AZD4635 monotherapy and AZD4635 combined with durvalumab in NSCLC (Arms F/G) and mCRPC (Arms I/J) in order to minimize bias.

Patients with CRC, excluding MSI high, will be enrolled to AZD4635 monotherapy (Arm K) and AZD4635 combined with durvalumab (Arm KD) in patients with CRC.

Some arms will have a mandatory biopsy subgroup to ensure sufficient tissue is collected to assess the mechanism of action in tissue without excluding patients with nonbiopsiable disease. Biopsies are optional in all other arms.

ELIGIBILITY:
Inclusion Criteria

1. Patient must consent to the study and provide a signed and dated written informed consent document prior to any study-specific procedures, sampling, or analyses.
2. Age ≥18 years
3. Weight ≥77 lbs (35 kg)
4. Availability of an archival tumor tissue sample. If archival tumor tissue is not available, then tissue from a fresh biopsy can be used.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 w/ no clinical deterioration over the prior 2 weeks (wks) and likely able to complete at least 9 wks of treatment.
6. Normotensive or well controlled blood pressure (systolic <150 and diastolic <90) w/ or without current anti-hypertensive treatment. If there is a diagnosis or history of hypertension, patient must have adequately controlled BP on antihypertensive medications as demonstrated by 2 BP measurements taken in the clinical setting by a medical professional within 1 week (wk) prior to enrollment. Patients on anti-hypertensive medication must be willing and able to check and record twice daily BP readings for a minimum of 3 wks.
7. Females should be using adequate contraceptive measures from the time of screening until 3 months after study discontinuation, should not be breast feeding and must have negative pregnancy test prior to the start of dosing, or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

   * Post-menopausal: defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
   * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not tubal ligation.
   * Women under 50 years-of-age will be considered postmenopausal if they have been amenorrheic for at least 12 months following the cessation of exogenous hormonal treatments, and have serum follicle-stimulating hormone and luteinizing hormone levels in the postmenopausal range for the institution.
8. Male patients should be willing to use barrier contraception for the duration of the study and for 3 months after treatment discontinuation.
9. Ability to swallow and retain oral medication.

Additional Inclusion Criteria for Phase 1a Arms AA and EA

1. Patients in Arms AA and EA must have metastatic prostate cancer w/ histological or cytological confirmation. Note: Patient may have bone only metastatic disease.

* Patients must be castrate-resistant (i.e. developed progression of metastases following surgical castration or during medical androgen ablation therapy). (Patients receiving medical castration therapy w/ gonadotropin-releasing hormone analogues should continue this treatment during this study.)
* Patients must have received prior treatment w/ at least one of the hormonal agents (abiraterone acetate, enzalutamide or apalutamide). Patients who received prior apalutamide will be allocated to abiraterone acetate (Arm AA). Note: Prior chemotherapy is allowed but not required.
* Patients must have evidence of disease progression.

Additional Inclusion Criteria for Phase 1a Arm CA

1. Patients in Arm CA must have a histologically/cytologically confirmed advanced solid tumor malignancy that has received and progressed on standard-of-care therapy(ies).

Additional Inclusion Criteria for Phase 1a Arms CB and CC

1. Patients in Arms CB and CC may have metastatic prostate cancer w/ histological or cytological confirmation:

   • Patient must be castrate-resistant (i.e., developed progression of metastases following surgical castration or during medical androgen ablation therapy). Patients receiving medical castration therapy with gonadotropin-releasing hormone analogues should continue this treatment during this study. Note: Patient with prostate cancer may have bone-only metastatic disease.

   • Patient must have-evidence of disease progression. Or

   • Patients in Cohort CB must have a histologically/cytologically confirmed advanced solid tumor malignancy that has received and progressed on standard-of-care therapy(ies).

   Or • Patients in Cohort CC should have a histologically/cytologically confirmed advanced solid tumor malignancy suitable for treatment with docetaxel.

   Additional Inclusion Criteria for Phase 1b

<!-- -->

1. Patients must have disease that is suitable for repeated measurement, either: a) at least one lesion that can be accurately assessed at baseline by computed tomography (CT), magnetic resonance imaging (MRI) or X-ray, that is suitable for repeated measurement (RECIST v1.1), or b) for patients with mCRPC (Arms I and J), patients must have measurable PSA above normal limits (per local ranges).
2. A minimum of 10 patients with mCRPC, CRC and 'Other' tumors will be required to have a site of disease that is safely accessible for biopsy (paired) upon enrollment. Accessible lesions are defined as those which are biopsiable (at screening) and amenable to repeat biopsy (after 2 wks of monotherapy), unless clinically contraindicated. In the case that the second sample is not taken, the patient will remain in the study and there will be no penalty or loss of benefit to the patient and they will not be excluded from other aspects of the study. The tumor-specific cohorts will be closely monitored to ensure the desired number of biopsiable patients are enrolled. The requirement for biopsies must be made clear to each patient at the time of initial approach by the Investigator.
3. For post immunotherapy patients with NSCLC (Arms F and G) all of the following must apply:

   * Patients must have advanced or metastatic NSCLC w/ histological or cytological confirmation. Patients with known EGFR-activating mutations or ALK rearrangements are excluded.
   * Patient must have previously received one (but no more than one) line of previous therapy w/ an anti-PD-1/PD-L1 mAb therapy either alone or in combination and have either progressed or responded and then stopped responding.
4. For other post-immunotherapy patients (Arm H) all of the following must apply:

   * Patients must have an immune checkpoint resistant malignancy (for example, RCC, head and neck carcinoma, or MSI high cancers which have approved settings for anti-PD1 treatment), confirmed histologically or cytologically.
   * Patients must have previously received at least one line (and not more than 2 lines) of previous therapy w/ an anti-PD-1/PD-L1 mAb therapy, either alone or in combination and have either progressed or responded and then stopped responding.
5. For immune checkpoint naïve CRPC patients (Arms I and J) all of the following must apply:

   • Patients must have metastatic prostate cancer w/ histological or cytological confirmation.
   * Patients must be castrate-resistant (i.e., developed progression of metastases following surgical castration or during medical androgen ablation therapy). Patients receiving medical castration therapy w/ gonadotropin-releasing hormone analog should continue this treatment during this study.
   * Patients must have previously received and progressed on standard-of-care therapy(ies).
   * Approximately 60 out of 80 patients w/ mCRPC enrolled must have measurable disease (approximately 30 out of 40 patients in each of the mCRPC arms I and J) that is suitable for repeated measurement (RECIST v1.1). Enrollment will be monitored to ensure the required number of patients with measurable disease enter the study.
6. For immune checkpoint naïve patients (Arms K and KD) all of the following must apply:

   * Patients must have immune checkpoint naïve histologically/cytologically confirmed advanced or metastatic colorectal carcinoma (CRC).
   * Patients must have previously received and progressed on at least 1 prior chemotherapy regimen.
7. For other immune checkpoint naïve tumor patients (Arm L) all of the following must apply:

   * Patients w/ other immune checkpoint naïve histologically/ cytologically confirmed advanced solid tumor type that has received and progressed on standard-of-care therapy(ies).

Exclusion Criteria

1. Treatment with any of the following:

   * Nitrosourea or mitomycin C within 6 wks of the first dose.
   * Any systemic anti-cancer chemotherapy, small molecule, biologic, or hormonal agent from a previous treatment regimen or clinical study within 21 days or 5 half-lives (whichever is shorter). At least 7 days must have elapsed between the last dose of such agent and the first dose of study drug. EXCEPTION: Androgen-deprivation therapy is recommended for patients w/ prostate cancer.
   * Enrollment into another therapeutic clinical trial. EXCEPTION: Patients are allowed to participate in investigational imaging or non-therapeutic studies.
   * Patient has had Rx or non-Rx drugs or other products known to be sensitive BCRP or OAT1 substrates or to be potent inhibitors/inducers of CYP1A2, which cannot be discontinued 2 wks prior to Day 1 of dosing and withheld throughout the study until 2 wks after the last dose of AZD4635.
   * Herbal preparations/medications are not allowed throughout the study, including but not limited to St. John's Wort, kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone, yohimbe, saw palmetto, and ginseng. Patients should stop using these herbal medications 7 days prior to the first dose of AZD4635.
   * Patient may not be assigned to abiraterone acetate arm (Arm AA) if co-administration of a strong CYP3A4 or a CYP2D6 substrate with a narrow therapeutic index is required during study treatment.
   * Patient may not be assigned to an enzalutamide arm (Arm EA) if co-administration of strong CYP2C8 inhibitor, strong or moderate CYP3A4 or CYP2C8 inducer, or CYP3A4, CYP2C9, and CYP2C19 substrates with a narrow therapeutic index is required during study treatment.
   * Ongoing treatment w/ Coumadin.
   * Concomitant medications w/ another A1R antagonist that would increase risk of seizure (e.g., theophylline or aminophylline).
   * AZD4635 in the present study (i.e., dosing w/ AZD4635 previously initiated in a different arm in this study), or prior therapy w/ AZD4635 or any other A2AR antagonist.
   * Ongoing corticosteroid use. NOTE: mCRPC patients assigned to an arm with abiraterone acetate (Arm AA) should take prednisone as prescribed for glucocorticoid replacement therapy and patients assigned to the docetaxel arm (Arm CC) should take prophylactic dexamethasone (or equivalent) to prevent severe hypersensitivity reactions.
   * Major surgery (excluding placement of vascular access) within 4 wks of the first dose of study treatment.
   * Radiotherapy w/ a wide field of radiation within 4 wks or radiotherapy w/ a limited field of radiation for palliation within 2 wks of the first dose of study treatment.
2. Patient w/ prior history of myocardial infarction, transient ischemic attack, or stroke within 3 months prior to the scheduled first dose of oleclumab treatment (Arm CB).
3. With the exception of alopecia, any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment must be discussed with the Medical Monitor.
4. History of seizures, central nervous system tumors or CNS metastasis. Due to the incidence of silent CNS metastases in patients with advanced NSCLC, such patients must undergo mandatory screening with brain MRI or CT scan to determine eligibility.
5. Significant mental illness in the 4-wk period preceding drug administration.
6. As judged by the investigator, any evidence of severe or uncontrolled systemic disease, including uncontrolled hypertension, active bleeding diatheses, or active infection, including hepatitis B, hepatitis C, and human immunodeficiency virus. Screening for chronic conditions is not required.
7. History or presence of another primary invasive malignancy except for:

   • Malignancy treated w/ curative intent and w/ no known active disease ≥2 years before the first dose of study drug and of low potential risk for recurrence.

   • Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.

   • Adequately treated carcinoma in situ without evidence of disease.

   • Localized non-invasive primary under surveillance.
8. Any of the following cardiac criteria:

   • Mean resting corrected QT interval (QTcF) >470 msec obtained from 3 ECGs.

   • Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECGs, e.g., complete left bundle branch block, third degree heart block.
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age, or any concomitant medication known to prolong the QT interval. Patients receiving a medication(s) known to prolong QT internval may be discussed w/ the Medical Monitor or Sponsor for study approval.
   * Ejection fraction <55% or less than the lower limit of normal of the institutional standard.
9. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

   • Absolute neutrophil count <1.5 x 10^9/L
   * Platelet count <100 x 10^9/L
   * Hemoglobin <90 g/L
   * ALT and/or AST >2.5 x the upper limit of normal (ULN) if no demonstrable liver metastases or >5 x ULN in the presence of liver metastases
   * Total bilirubin >1.5 x ULN
   * Creatinine >1.5 x ULN concurrent with creatinine clearance <50 mL/min
10. Refractory nausea and vomiting, chronic gastrointestinal diseases, or previous significant bowel resection that would preclude adequate absorption of AZD4635.
11. Any patient w/ open oral ulceration(s) should avoid dosing with AZD4635 oral suspension.
12. Patients w/ severe hepatic impairment (Child-Pugh Class C) are not permitted to enroll in the mCRPC plus hormone arms containing abiraterone acetate.
13. Organ transplant that requires the use of immunosuppressive treatment.
14. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g. colitis, Crohn's disease], diverticulitis, celiac disease, systemic lupus erythematous, Wegner's syndrome, myasthenia gravis, Grave's disease, rheumatoid arthritis, hypophysitis, uveitis, autoimmune pneumonitis, autoimmune nephritis or nephropathy, etc.) within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

    * Vitiligo or alopecia.
    * Hypothyroidism (e.g., following Hashimoto's disease) stable on hormone replacement.
    * Psoriasis or eczema not requiring systemic treatment.
15. Patients w/ prior ≥Grade 3, serious, or life threatening immune-mediated reactions following prior anti-PD-1 or other immune-oncology therapies.
16. History of hypersensitivity to AZD4635 or drugs w/ a similar chemical structure or class to AZD4635.
17. Judgment by the Investigator or the Medical Monitor that the patient should not participate in the study if the patient is unlikely to comply w/ study procedures, restrictions, and/or requirements.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2016-06-17 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
The incidence of Dose-Limiting Toxicities (DLTs) in patients receiving AZD4635 monotherapy orally. | 3 weeks (One Cycle)
  A Bayesian Logistic Regression Model (BLRM) based approach will be used to identify the set of AZD4635 doses where the incidence of DLTs is no larger than 33%. In each arm, up to 3 patients will be initially assessed. The dose will be escalated to the next higher dose level if all 3 patients in the previous dose level complete the DLT evaluation period without a DLT. Following the first DLT, the BLRM model will be run and the output made available to the safety review committee (SRC) to guide further dosing decisions. Each dose cohort will include a maximum of 6 patients.
The incidence of Dose-Limiting Toxicities (DLTs) in patients receiving AZD4635 in combination with durvalumab. | 7 weeks (Including Cycle 0)
  A Bayesian Logistic Regression Model (BLRM) based approach will be used to identify the set of AZD4635 doses where the incidence of DLTs is no larger than 33%. In each arm, up to 3 patients will be initially assessed. The dose will be escalated to the next higher dose level if all 3 patients in the previous dose level complete the DLT evaluation period without a DLT. Following the first DLT, the BLRM model will be run and the output made available to the safety review committee (SRC) to guide further dosing decisions. Each dose cohort will include a maximum of 6 patients.
The incidence of Dose-Limiting Toxicities (DLTs) in patients receiving AZD4635 in combination with either abiraterone acetate or enzalutamide. | 21 days (Cycle 1)
  The starting dose of AZD4635 is 50 mg PO QD. Escalations of AZD4635 will be made based on emerging data, including nonclinical or clinical evidence, and assessment by the Safety Review Committee (SRC). Each dose cohort will include a maximum of 6 evaluable patients. An additional 6 patients will be treated at selected dose(s) to obtain further the safety, tolerability, and PK.
The incidence of adverse events | Patients will be followed for either 21 days in Cycles 1 and 2 or 28 days in Cycles 3 and beyond to determine the incidence of adverse events.
  Safety and tolerability will be assessed in monotherapy and combination cohorts by determining the incidence of adverse events, including abnormal laboratory results, physical examination findings, vital signs, and urinalysis.

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) of AZD4635 after single-dose administration in Cycle 0 | Samples will be collected at pre-specified time points for up to one-week following a single-dose of AZD4635 (Cycle 0). The multiple-dose PK sampling will commence with Cycle 1 Day 1.
  The plasma concentration of AZD4635 will be determined by inspection of the concentration-time profile. Intensive pharmacokinetic sampling with matched ECGs is required in Phase 1a and in NSCLC Cohorts and mCRPC Cohorts in the monotherapy portion of the study. After the pharmacokinetic profile has been sufficiently characterised, sample collection in the mCRPC and NSCLC expansion cohorts may be limited to coincide with ECG-matched time points in patients being newly enrolled. Sparse sample collections are required from patients in CRC, Post-IO Other, and IO-Naïve Other cohorts.
Time to peak plasma concentration (tmax) of AZD4635 after single-dose administration in Cycle 0 | Samples will be collected at pre-specified time points for up to one-week following a single-dose of AZD4635 (Cycle 0). The multiple-dose PK sampling will commence with Cycle 1 Day 1.
  The plasma concentration of AZD4635 will be determined by inspection of the concentration-time profile. Intensive pharmacokinetic sampling with matched ECGs is required in Phase 1a and in NSCLC Cohorts and mCRPC Cohorts in the monotherapy portion of the study. After the pharmacokinetic profile has been sufficiently characterised, sample collection in the mCRPC and NSCLC expansion cohorts may be limited to coincide with ECG-matched time points in patients being newly enrolled. Sparse sample collections are required from patients in CRC, Post-IO Other, and IO-Naïve Other cohorts.
Terminal elimination rate constant (λz) of AZD4635 after single-dose administration in Cycle 0 | Samples will be collected at pre-specified time points for up to one-week following a single-dose of AZD4635 (Cycle 0). The multiple-dose PK sampling will commence with Cycle 1 Day 1.
  The plasma concentration of AZD4635 will be determined by inspection of the concentration-time profile. Intensive pharmacokinetic sampling with matched ECGs is required in Phase 1a and in NSCLC Cohorts and mCRPC Cohorts in the monotherapy portion of the study. After the pharmacokinetic profile has been sufficiently characterised, sample collection in the mCRPC and NSCLC expansion cohorts may be limited to coincide with ECG-matched time points in patients being newly enrolled. Sparse sample collections are required from patients in CRC, Post-IO Other, and IO-Naïve Other cohorts.
Terminal elimination half-life (t½λz) of AZD4635 after single-dose administration in Cycle 0 | Samples will be collected at pre-specified time points for up to one-week following a single-dose of AZD4635 (Cycle 0). The multiple-dose PK sampling will commence with Cycle 1 Day 1.
  The plasma concentration of AZD4635 will be determined by inspection of the concentration-time profile. Intensive pharmacokinetic sampling with matched ECGs is required in Phase 1a and in NSCLC Cohorts and mCRPC Cohorts in the monotherapy portion of the study. After the pharmacokinetic profile has been sufficiently characterised, sample collection in the mCRPC and NSCLC expansion cohorts may be limited to coincide with ECG-matched time points in patients being newly enrolled. Sparse sample collections are required from patients in CRC, Post-IO Other, and IO-Naïve Other cohorts.
Area under the plasma concentration-time curve following single dose administration of AZD4635 in Cycle 0 | Samples will be collected at pre-specified time points for up to one-week following a single-dose of AZD4635 (Cycle 0). The multiple-dose PK sampling will commence with Cycle 1 Day 1
  The plasma concentration of AZD4635 will be determined by inspection of the concentration-time profile. Intensive pharmacokinetic sampling with matched ECGs is required in Phase 1a and in NSCLC Cohorts and mCRPC Cohorts in the monotherapy portion of the study. After the pharmacokinetic profile has been sufficiently characterised, sample collection in the mCRPC and NSCLC expansion cohorts may be limited to coincide with ECG-matched time points in patients being newly enrolled. Sparse sample collections are required from patients in CRC, Post-IO Other, and IO-Naïve Other cohorts.
Apparent plasma clearance (CL/F) after single-dose administration of AZD4635 in Cycle 0 | Samples will be collected at pre-specified time points for up to one-week following a single-dose of AZD4635 (Cycle 0). The multiple-dose PK sampling will commence with Cycle 1 Day 1.
  The plasma concentration of AZD4635 will be determined by inspection of the concentration-time profile. Intensive pharmacokinetic sampling with matched ECGs is required in Phase 1a and in NSCLC Cohorts and mCRPC Cohorts in the monotherapy portion of the study. After the pharmacokinetic profile has been sufficiently characterised, sample collection in the mCRPC and NSCLC expansion cohorts may be limited to coincide with ECG-matched time points in patients being newly enrolled. Sparse sample collections are required from patients in CRC, Post-IO Other, and IO-Naïve Other cohorts.
Apparent volume of distribution (Vz/F) after single-dose administration of AZD4635 in Cycle 0 | Samples will be collected at pre-specified time points for up to one-week following a single-dose of AZD4635 (Cycle 0). The multiple-dose PK sampling will commence with Cycle 1 Day 1.
  The plasma concentration of AZD4635 will be determined by inspection of the concentration-time profile. Intensive pharmacokinetic sampling with matched ECGs is required in Phase 1a and in NSCLC Cohorts and mCRPC Cohorts in the monotherapy portion of the study. After the pharmacokinetic profile has been sufficiently characterised, sample collection in the mCRPC and NSCLC expansion cohorts may be limited to coincide with ECG-matched time points in patients being newly enrolled. Sparse sample collections are required from patients in CRC, Post-IO Other, and IO-Naïve Other cohorts.
Mean residence time (MRT) of AZD4635 after single-dose administration in Cycle 0 | Samples will be collected at pre-specified time points for up to one-week following a single-dose of AZD4635 (Cycle 0). The multiple-dose PK sampling will commence with Cycle 1 Day 1.
  The plasma concentration of AZD4635 will be determined by inspection of the concentration-time profile. Intensive pharmacokinetic sampling with matched ECGs is required in Phase 1a and in NSCLC Cohorts and mCRPC Cohorts in the monotherapy portion of the study. After the pharmacokinetic profile has been sufficiently characterised, sample collection in the mCRPC and NSCLC expansion cohorts may be limited to coincide with ECG-matched time points in patients being newly enrolled. Sparse sample collections are required from patients in CRC, Post-IO Other, and IO-Naïve Other cohorts.
Renal clearance (CLR) of AZD4635 after single-dose administration in Cycle 0 | Samples will be collected at pre-specified time points for up to one-week following a single-dose of AZD4635 (Cycle 0). The multiple-dose PK sampling will commence with Cycle 1 Day 1.
  The plasma concentration of AZD4635 will be determined by inspection of the concentration-time profile. Intensive pharmacokinetic sampling with matched ECGs is required in Phase 1a and in NSCLC Cohorts and mCRPC Cohorts in the monotherapy portion of the study. After the pharmacokinetic profile has been sufficiently characterised, sample collection in the mCRPC and NSCLC expansion cohorts may be limited to coincide with ECG-matched time points in patients being newly enrolled. Sparse sample collections are required from patients in CRC, Post-IO Other, and IO-Naïve Other cohorts.
Amount of AZD4635 excreted unchanged in urine (Ae) after single-dose administration in Cycle 0 | Urine will be collected and pooled at specific intervals: pre-dose (spot urine), 0 to 4 hours, 4 to 8 hours, and 8 to 24 hours.
  The amount of AZD4635 (and metabolites) in urine will be determined in all patients. Pooled collections of urine 0 to 4 hours post dose, 4 to 8 hours post dose, and 8 to 24 hours post dose. Patients will collect all urine at home and bring the 8 to 24 hour pooled collection to the clinic. The total volume of each pooled sample will be recorded after which a 10 mL aliquot will be taken for analysis.
Fraction of AZD4635 excreted unchanged in urine (fe) after single-dose administration in Cycle 0 | Urine will be collected and pooled at specific intervals: pre-dose (spot urine), 0 to 4 hours, 4 to 8 hours, and 8 to 24 hours.
  The amount of AZD4635 (and metabolites) in urine will be determined in all patients. Pooled collections of urine 0 to 4 hours post dose, 4 to 8 hours post dose, and 8 to 24 hours post dose. Patients will collect all urine at home and bring the 8 to 24 hour pooled collection to the clinic. The total volume of each pooled sample will be recorded after which a 10 mL aliquot will be taken for analysis.
Peak plasma concentration of AZD4635 at steady state (Cmax, ss) following multiple-doses on Cycle 1 Day 15 in monotherapy arms and Cycle 1 Day 1 and Cycle 3 Day 15 in combination therapy arms. | Samples will be collected at pre-specified time points in the multiple-dose portion of the study beginning with Cycle 1 Day 1. Sampling be done on 1 of 3 schedules: i) Intensive sampling, ii) ECG-matched sampling, or iii) Sparse sampling.
  The plasma concentration of AZD4635 will be determined by inspection of the concentration-time profile. Intensive pharmacokinetic sampling with matched ECGs is required in Phase 1a and in NSCLC Cohorts and mCRPC Cohorts in the monotherapy portion of the study. After the pharmacokinetic profile has been sufficiently characterised, sample collection in the mCRPC and NSCLC expansion cohorts may be limited to coincide with ECG-matched time points in patients being newly enrolled. Sparse sample collections are required from patients in CRC, Post-IO Other, and IO-Naïve Other cohorts.
Time to peak plasma concentration of AZD4635 at steady state (tmax, ss) following multiple-doses on Cycle 1 Day 15 in monotherapy arms and Cycle 1 Day 1 and Cycle 3 Day 15 in combination therapy arms. | Samples will be collected at pre-specified time points in the multiple-dose portion of the study beginning with Cycle 1 Day 1. Sampling be done on 1 of 3 schedules: i) Intensive sampling, ii) ECG-matched sampling, or iii) Sparse sampling.
  The plasma concentration of AZD4635 will be determined by inspection of the concentration-time profile. Intensive pharmacokinetic sampling with matched ECGs is required in Phase 1a and in NSCLC Cohorts and mCRPC Cohorts in the monotherapy portion of the study. After the pharmacokinetic profile has been sufficiently characterised, sample collection in the mCRPC and NSCLC expansion cohorts may be limited to coincide with ECG-matched time points in patients being newly enrolled. Sparse sample collections are required from patients in CRC, Post-IO Other, and IO-Naïve Other cohorts.
Minimum plasma concentration of AZD4635 at steady state (Cmin, ss) following multiple-doses on Cycle 1 Day 15 in monotherapy arms and Cycle 1 Day 1 and Cycle 3 Day 15 in combination therapy arms. | Samples will be collected at pre-specified time points in the multiple-dose portion of the study beginning with Cycle 1 Day 1. Sampling be done on 1 of 3 schedules: i) Intensive sampling, ii) ECG-matched sampling, or iii) Sparse sampling.
  The plasma concentration of AZD4635 will be determined by inspection of the concentration-time profile. Intensive pharmacokinetic sampling with matched ECGs is required in Phase 1a and in NSCLC Cohorts and mCRPC Cohorts in the monotherapy portion of the study. After the pharmacokinetic profile has been sufficiently characterised, sample collection in the mCRPC and NSCLC expansion cohorts may be limited to coincide with ECG-matched time points in patients being newly enrolled. Sparse sample collections are required from patients in CRC, Post-IO Other, and IO-Naïve Other cohorts.
Area under the plasma concentration-time curve within the dosing interval (AUCtau) following multiple-doses on Cycle 1 Day 15 in monotherapy arms and Cycle 1 Day 1 and Cycle 3 Day 15 in combination therapy arms. | Samples will be collected at pre-specified time points in the multiple-dose portion of the study beginning with Cycle 1 Day 1. Sampling be done on 1 of 3 schedules: i) Intensive sampling, ii) ECG-matched sampling, or iii) Sparse sampling.
  The plasma concentration of AZD4635 will be determined by inspection of the concentration-time profile. Intensive pharmacokinetic sampling with matched ECGs is required in Phase 1a and in NSCLC Cohorts and mCRPC Cohorts in the monotherapy portion of the study. After the pharmacokinetic profile has been sufficiently characterised, sample collection in the mCRPC and NSCLC expansion cohorts may be limited to coincide with ECG-matched time points in patients being newly enrolled. Sparse sample collections are required from patients in CRC, Post-IO Other, and IO-Naïve Other cohorts.
Apparent plasma clearance at steady state (CLss/F) following multiple-doses on Cycle 1 Day 15 in monotherapy arms and Cycle 1 Day 1 and Cycle 3 Day 15 in combination therapy arms. | Samples will be collected at pre-specified time points in the multiple-dose portion of the study beginning with Cycle 1 Day 1. Sampling be done on 1 of 3 schedules: i) Intensive sampling, ii) ECG-matched sampling, or iii) Sparse sampling.
  The plasma concentration of AZD4635 will be determined by inspection of the concentration-time profile. Intensive pharmacokinetic sampling with matched ECGs is required in Phase 1a and in NSCLC Cohorts and mCRPC Cohorts in the monotherapy portion of the study. After the pharmacokinetic profile has been sufficiently characterised, sample collection in the mCRPC and NSCLC expansion cohorts may be limited to coincide with ECG-matched time points in patients being newly enrolled. Sparse sample collections are required from patients in CRC, Post-IO Other, and IO-Naïve Other cohorts.
Extent of accumulation of AZD4635 (Rac) after multiple dosing | Samples will be collected at pre-specified time points in the multiple-dose portion of the study beginning with Cycle 1 Day 1. Sampling will be done on 1 of 3 schedules: i) Intensive sampling, ii) ECG-matched sampling, or iii) Sparse sampling.
  The plasma concentration of AZD4635 will be determined by inspection of the concentration-time profile. Intensive pharmacokinetic sampling with matched ECGs is required in Phase 1a and in NSCLC Cohorts and mCRPC Cohorts in the monotherapy portion of the study. After the pharmacokinetic profile has been sufficiently characterised, sample collection in the mCRPC and NSCLC expansion cohorts may be limited to coincide with ECG-matched time points in patients being newly enrolled. Sparse sample collections are required from patients in CRC, Post-IO Other, and IO-Naïve Other cohorts.
Time dependency of AZD4635 pharmacokinetic parameters (TCP) after multiple dosing. | Samples will be collected at pre-specified time points in the multiple-dose portion of the study beginning with Cycle 1 Day 1. Sampling will be done on 1 of 3 schedules: i) Intensive sampling, ii) ECG-matched sampling, or iii) Sparse sampling.
  The plasma concentration of AZD4635 will be determined by inspection of the concentration-time profile. Intensive pharmacokinetic sampling with matched ECGs is required in Phase 1a and in NSCLC Cohorts and mCRPC Cohorts in the monotherapy portion of the study. After the pharmacokinetic profile has been sufficiently characterised, sample collection in the mCRPC and NSCLC expansion cohorts may be limited to coincide with ECG-matched time points in patients being newly enrolled. Sparse sample collections are required from patients in CRC, Post-IO Other, and IO-Naïve Other cohorts.
The concentration of durvalumab and anti-drug antibody in plasma when given in combination with AZD4635 | Preinfusion and end of infusion on Day 1 of Cycles 2 and 5. Preinfusion of Day 1 of Cycles 3 and 8 and 90-days after the last dose of durvalumab.
  Plasma concentration of durvalumab and anti-drug antibody will be determined by inspection of the concentration-time profile. The date and time of collection of each sample will be recorded.
The effect of AZD4635 on QTc interval | In screening and on Days 1, 2 and 15 in Cycle 1, Day 1 of each cycle thereafter, and at the end of treatment and at each progression-free follow-up visit.
  Twelve-lead ECGs will be obtained after the patient has been resting supine for at least 10 minutes. For each time point 3 ECG recordings should be taken at about 2- to 5 minute intervals.
Tumour Response | Tumour response will be assessed 6 weeks after the start of treatment and then every 8 weeks; after 18 months, assessments will be every 12 weeks.
  Categorization of objective tumour response assessment will be based on the RECIST Version 1.1 guidelines for response (CR (complete response), PR (partial response), SD (stable disease), and PD (progressive disease).
  For patients who only have non-measurable disease at baseline, categorization of objective tumour response assessment will be based on the RECIST Version 1.1 guideline for response for non-target lesions (NTLs): CR, PD, and Non CR/Non PD.
Progression free survival | Patients will be restaged after 6 weeks (+/- 7 days) and every 8 weeks (+/- 7 days) thereafter, at the end of treatment visit if required, and at progression free follow up visits if they discontinue study treatment prior to progression.
  Progression free survival is defined as the time interval from the first dose of AZD4635 until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from study treatment. Subjects who have not progressed or died at the time of analysis will be censored at the time of the last evaluable RECIST assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Bendell, MD, Study Chair — SCRI Development Innovations, LLC
Locations (17):
- United States (17):
  - Research Site, Fayetteville, Arkansas
  - Research Site, Fresno, California
  - Research Site, Denver, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Daytona Beach, Florida
  - Research Site, Lecanto, Florida
  - Research Site, North Port, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Decatur, Illinois
  - Research Site, Las Vegas, Nevada
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8730C00001&attachmentIdentifier=3d8cb6f0-b036-4681-baf4-509f928ead35&fileName=d8730c00001-study-synopsis-Redacted.pdf&versionIdentifier=